CLINICAL TRIAL: NCT06783699
Title: Comparisons of Urodynamic and Clinical Findings Between Those Positive and Negative sUPP in Women With Urodynamic Stress Incontinence
Brief Title: Comparison Between Positive and Negative sUPP
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202406048RINC
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-06

CONDITIONS: Urodynamic Stress Incontinence
Keywords: Urodynamic stress incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive sUPP: Involuntary urine leak during cough stress test in urethral pressure profile
- Negative sUPP: No urine leak during cough stress test in urethral pressure profile

SUMMARY:
Urodynamic stress incontinence is a prevalent condition among women, characterized by involuntary urine leakage during activities that increase intra-abdominal pressure, such as coughing, sneezing, or physical exertion. Stress urethral pressure profile measurement is an important diagnostic tool used during urodynamic studies to assess urethral function. In some women with urodynamic stress incontinence, involuntary urine leakage occurs during this measurement, yet the clinical and urodynamic significance of this leakage remains unclear. This study aims to elucidate the differences in clinical and urodynamic findings between women with urodynamic stress incontinence who experience involuntary urine leakage during stress urethral pressure profile measurement and those who do not. Between July 2009 and December 2023, a total of 481 women with urodynamic stress incontinence were included and divided into positive and negative sUPP groups. The medical records, including urodynamic study, 3-day bladder dairy and questionnaires regarding lower urinary tract symptoms were reviewed.

DETAILED DESCRIPTION:
Hypothesis / aims of study Involuntary urine leakage has been observed during stress urethral pressure measurement in women with urodynamic stress incontinence (USI). However, to our knowledge, its clinical significance and urodynamic association remained undetermined. Therefore, the objective of this study is to elucidate the above differences between those with versus without involuntary urine leakage during the measurement of stress urethral pressure in women with USI.

Study design, materials and methods Between July 2009 and December 2023, medical records, including urodynamic data, bladder dairy data and questionnaires, including patient perception of bladder condition (PPBC), urgency severity scale (USS), overactive bladder symptom score (OABSS), urogenital distress inventory (UDI-6), incontinence impact questionnaire (IIQ-7), and King's Health Questionnaire (KHQ), of all women with USI were reviewed to see if there was any involuntary leakage of urine during stress urethral pressure measurement.

STATA software was used for statistical analysis. The Wilcoxon rank sum test or the Chi-square test were used for statistical analysis, as appropriate. A p < 0.05 was considered statistically significant. Linear regression analysis was also performed with an adjustment of overactive bladder syndrome (OAB) to elucidate the real clinical and urodynamic associations about the leak during stress urethral pressure measurement.

ELIGIBILITY:
Inclusion Criteria:

* >20 y/o
* Women with lower urinary tract symptoms
* Received urodynamic stress incontinence and was diagnosed with urodynamic stress incontinence

Exclusion Criteria:

* Women who are pregnant
* With chronic pelvic inflammatory disease

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged more than 20-year-old with lower urinary tract symptoms underwent urodynamic study and were diagnosed with urodynamic stress incontinence.
Sampling Method: Non-Probability Sample
Enrollment: 481 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence in bladder diary | Between July 2009 and December 2023
  Subjective urinary incontinence described in bladder diary

SECONDARY OUTCOMES:
Pad weight | Between July 2009 and December 2023
  Pad weight in pad test

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, M.D. Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Data will be shared under request.

REFERENCES:
- [Result] Wu PC, Hsiao SM, Lin HH. Prevalence and predictors of nocturnal polyuria in females with overactive bladder syndrome. World J Urol. 2022 Feb;40(2):519-527. doi: 10.1007/s00345-021-03865-5. Epub 2021 Nov 11. PMID 34762173
- [Result] Hsiao SM, Wu PC, Chang TC, Chen CH, Lin HH. Urodynamic and Bladder Diary Factors Predict Overactive Bladder-wet in Women: A Comparison With Overactive Bladder-dry. Int Neurourol J. 2019 Mar;23(1):69-74. doi: 10.5213/inj.1836212.106. Epub 2019 Mar 31. PMID 30943696
- [Result] Hsiao SM, Hsiao CF, Chen CH, Chang TC, Wu WY, Lin HH. Evaluation of bladder diary parameters based on correlation with the volume at strong desire to void in filling cystometry. PLoS One. 2013 Jul 29;8(7):e69946. doi: 10.1371/journal.pone.0069946. Print 2013. PMID 23922866
- [Result] Rosier PFWM, Schaefer W, Lose G, Goldman HB, Guralnick M, Eustice S, Dickinson T, Hashim H. International Continence Society Good Urodynamic Practices and Terms 2016: Urodynamics, uroflowmetry, cystometry, and pressure-flow study. Neurourol Urodyn. 2017 Jun;36(5):1243-1260. doi: 10.1002/nau.23124. Epub 2016 Dec 5. PMID 27917521
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278